CLINICAL TRIAL: NCT00277277
Title: Telehealth Delivery of a Weight Loss Program in Diabetes
Brief Title: In-Home Weight Loss Program for Adults With Type 2 Diabetes Delivered by Interactive Cable Television Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R21 EG002311-02
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Telemedicine; Biobehavioral weight loss program; Body Mass Index; Blood Glucose; Diabetes Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Healthium

SUMMARY:
The majority of patients with Type 2 Diabetes are obese and weight loss is known to improve diabetes outcomes and reduce the need for anti-diabetic medical. This 8-week Telehealth study will compare the effects of standard weight loss advice given in a clinic setting to weight loss advice delivered in the home using an interactive cable television technology called Healthium.

DETAILED DESCRIPTION:
The majority of patients with Type 2 Diabetes are obese and weight loss is known to improve diabetes outcomes and reduce the need for anti-diabetic medical. The overall goal of this study is to explore the human engineering issues of a home (non-clinical) telehealth system, Healthium, utilizing an interactive television system over a broadband connection.

The study seeks to demonstrate a convenient, intuitive and inexpensive way to conduct large-scale interventions related to obesity and nutrition. This could lead to a viable public health care initiative for prevention of chronic diseases such as diabetes. The specific aims to be addressed are Aim #1: To transfer a successful internet-based weight loss program onto the Healthium interactive platform and further develop the intervention for use in patients with Type 2 diabetes. Aim #2: To conduct focus groups to determine consumer acceptability of the convenience and intuitiveness of the Healthium interface. Aim #3: To perform a pilot study in patients with Type 2 diabetes to determine whether the Healthium interface improves weight loss and diabetes outcomes relative to standard clinic-based treatment over a period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria: Clinical Diagnosis of TYpe 2 Diabetes, Body Mass Index 25-35; Ability to read at 8th grade level, have a working television set in the household, be willing to complete daily exercise and diet logs for the 8-233k study; be willing to attend at least 3 clinic visits; Under care of physician for diabetes -

Exclusion Criteria: Evidence of cardiac, renal, or other endocrine diseases; clinical evidence of a substance abuse or mental illness; pregnancy or anticipated pregnancy; breastfeeding; excessive alcohol consumption; anticipated major lifestyle changes

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2004-08; Study Completion 2005-09

PRIMARY OUTCOMES:
Body weight at 8 weeks; Body Mass Index at 8 weeks; Diabetes outcomes at 8 weeks

SECONDARY OUTCOMES:
Hip/waist circumference at 8 weeks; Energy and nutrient intake at 8 weeks; Physical activity at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lovejoy, PhD, Principal Investigator — Bastyr University
Locations (1):
- Bastyr Center for Natural Health, Seattle, Washington, United States

REFERENCES:
- [Background] Ahring KK, Ahring JP, Joyce C, Farid NR. Telephone modem access improves diabetes control in those with insulin-requiring diabetes. Diabetes Care. 1992 Aug;15(8):971-5. doi: 10.2337/diacare.15.8.971. PMID 1505329
- [Background] Barnard RJ, Jung T, Inkeles SB. Diet and exercise in the treatment of NIDDM. The need for early emphasis. Diabetes Care. 1994 Dec;17(12):1469-72. doi: 10.2337/diacare.17.12.1469. PMID 7882819
- [Background] Currell R, Urquhart C, Wainwright P, Lewis R. Telemedicine versus face to face patient care: effects on professional practice and health care outcomes. Nurs Times. 2001 Aug 30-Sep 5;97(35):35. No abstract available. PMID 11957594
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Friedman RH, Kazis LE, Jette A, Smith MB, Stollerman J, Torgerson J, Carey K. A telecommunications system for monitoring and counseling patients with hypertension. Impact on medication adherence and blood pressure control. Am J Hypertens. 1996 Apr;9(4 Pt 1):285-92. doi: 10.1016/0895-7061(95)00353-3. PMID 8722429
- [Background] Harvey-Berino J, Pintauro S, Buzzell P, DiGiulio M, Casey Gold B, Moldovan C, Ramirez E. Does using the Internet facilitate the maintenance of weight loss? Int J Obes Relat Metab Disord. 2002 Sep;26(9):1254-60. doi: 10.1038/sj.ijo.0802051. PMID 12187404
- [Background] Hersh WR, Wallace JA, Patterson PK, Shapiro SE, Kraemer DF, Eilers GM, Chan BK, Greenlick MR, Helfand M. Telemedicine for the Medicare population: pediatric, obstetric, and clinician-indirect home interventions. Evid Rep Technol Assess (Summ). 2001 Aug;(24 Suppl):1-32. PMID 11569328
- [Background] Meyers AW, Graves TJ, Whelan JP, Barclay DR. An evaluation of a television-delivered behavioral weight loss program: are the ratings acceptable? J Consult Clin Psychol. 1996 Feb;64(1):172-8. doi: 10.1037//0022-006x.64.1.172. PMID 8907097
- [Background] Mokdad AH, Ford ES, Bowman BA, Nelson DE, Engelgau MM, Vinicor F, Marks JS. Diabetes trends in the U.S.: 1990-1998. Diabetes Care. 2000 Sep;23(9):1278-83. doi: 10.2337/diacare.23.9.1278. PMID 10977060
- [Background] Starren J, Hripcsak G, Sengupta S, Abbruscato CR, Knudson PE, Weinstock RS, Shea S. Columbia University's Informatics for Diabetes Education and Telemedicine (IDEATel) project: technical implementation. J Am Med Inform Assoc. 2002 Jan-Feb;9(1):25-36. doi: 10.1136/jamia.2002.0090025. PMID 11751801
- [Background] Shea S, Starren J, Weinstock RS, Knudson PE, Teresi J, Holmes D, Palmas W, Field L, Goland R, Tuck C, Hripcsak G, Capps L, Liss D. Columbia University's Informatics for Diabetes Education and Telemedicine (IDEATel) Project: rationale and design. J Am Med Inform Assoc. 2002 Jan-Feb;9(1):49-62. doi: 10.1136/jamia.2002.0090049. PMID 11751803
- [Background] Tate DF, Wing RR, Winett RA. Using Internet technology to deliver a behavioral weight loss program. JAMA. 2001 Mar 7;285(9):1172-7. doi: 10.1001/jama.285.9.1172. PMID 11231746
- [Background] Watts NB, Spanheimer RG, DiGirolamo M, Gebhart SS, Musey VC, Siddiq YK, Phillips LS. Prediction of glucose response to weight loss in patients with non-insulin-dependent diabetes mellitus. Arch Intern Med. 1990 Apr;150(4):803-6. PMID 2327840
- [Background] Wing RR, Shoemaker M, Marcus MD, McDermott M, Gooding W. Variables associated with weight loss and improvements in glycemic control in type II diabetic patients in behavioral weight control programs. Int J Obes. 1990 Jun;14(6):495-503. PMID 2401586
- [Background] Yamanouchi K, Shinozaki T, Chikada K, Nishikawa T, Ito K, Shimizu S, Ozawa N, Suzuki Y, Maeno H, Kato K, et al. Daily walking combined with diet therapy is a useful means for obese NIDDM patients not only to reduce body weight but also to improve insulin sensitivity. Diabetes Care. 1995 Jun;18(6):775-8. doi: 10.2337/diacare.18.6.775. PMID 7555502